CLINICAL TRIAL: NCT02804477
Title: Validation and Assessment of Patient Adherence to Opioids for Cancer Pain Using MMAS 8 Questionnaire in Pain Clinic
Brief Title: Validation and Assessment of Patient Adherence to Opioids for Cancer Pain Using MMAS 8 Pain Clinic
Status: Completed | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Parmanand Jain, Professor, Tata Memorial Centre
Other Study IDs: TataMC 1680
Record Dates: First submitted 2016-06-13; First posted 2016-06-17 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Chronic Cancer Pain
Keywords: adherence; opioid; MMAS 8, morisky medication adherence scale; validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims at finding degree of adherence of patients to their chronic pain medication prescriptions containing opioid e.g. Morphine, using Morisky Medication Adherence Scale 8, self- reported questionnaire. Also relationship of various demographic, disease related and opioid related factors to medication adherence.

DETAILED DESCRIPTION:
After institutional review board approval, a Pilot study including 30 patients will be conducted to validate Morisky Medication Adherence Scale 8 to validate the questionnaire for cross cultural variation. The data collected will be analyzed and result will be submitted to institutional review board for approval to conduct the parent study. Following the above approval, all adult patients , more than 18 yrs. of age, who are on a strong opioid for their chronic cancer pain, taken prescription from pain clinic at least once in past, who are able to understand and communicate Hindi will be invited to participate in the study. Each patient will be verbally asked about their medication and same will be confirmed by their previous medical records. An informed written consent will be obtained. Data will be collected by PI or co-investigator after obtaining written consent at Pain clinic(general and private) of Tata Memorial Hospital. Fund for purchasing the copyright to use the Hindi translation of Morisky Medication Adherence Scale 8, was provided by the department of Anesthesia Account, Tata Memorial Hospital, after due permission obtained from, Director Tata Memorial Center and Head of the department of Anesthesiology, critical care and pain, Tata Memorial Center. The precise scoring and permission to use the Hindi translation of the scale has been obtained from the developer. For income we will be considering private and general category of the patients respectively.Data will be analyzed using International Business machines software package for statistical analysis version 20.0.Pilot study data will be analyzed applying tests as internal consistency (Cronbach's alfa), Test retest variability and factor analysis.For parent study in the uni-variate analysis all variables listed above will consecutively tested for significant associations with ''good adherence'' as the outcome variable. Chi-square tests and Student's t-tests will used for categorical and continuous variables, respectively. All variables will be unconditionally entered into a binary logistic multi variate analysis. All p values #0.05 will regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. All adult patients > 18 yrs. of age
2. Patients suffering from chronic pain of any type and severity 3. On opioid i.e. Morphine, taken prescription at least once 4. Who can understand and communicate Hindi

Exclusion Criteria:

1. Refusal of consent
2. Paediatric patients
3. Patients who cannot understand or communicate Hindi

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting to pain clinic( private and general) will be screened and enrolled according to inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
validation and assessment of adherence to opioids for chronic cancer pain in pain clinic using Morisky medication adherence scale 8 | six months
  to do a pilot study comprising of 30 patients for cross cultural validation of Morisky medication adherence questionnaire , if it gets validated then assessment of adherence of patients suffering from chronic cancer pain to opioids.

SECONDARY OUTCOMES:
relationship of adherence to opioids with demographic characteristics | six months

CONTACTS AND LOCATIONS:
Overall Officials: Parmanand Jain, MD, Principal Investigator — Professor; charushree E jibhkate, Junior resident, Study Chair — Junior resident
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Larue F, Colleau SM, Brasseur L, Cleeland CS. Multicentre study of cancer pain and its treatment in France. BMJ. 1995 Apr 22;310(6986):1034-7. doi: 10.1136/bmj.310.6986.1034. PMID 7728056
- [Background] van den Beuken-van Everdingen MH, de Rijke JM, Kessels AG, Schouten HC, van Kleef M, Patijn J. Prevalence of pain in patients with cancer: a systematic review of the past 40 years. Ann Oncol. 2007 Sep;18(9):1437-49. doi: 10.1093/annonc/mdm056. Epub 2007 Mar 12. PMID 17355955
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Krousel-Wood M, Hyre A, Muntner P, Morisky D. Methods to improve medication adherence in patients with hypertension: current status and future directions. Curr Opin Cardiol. 2005 Jul;20(4):296-300. doi: 10.1097/01.hco.0000166597.52335.23. PMID 15956826